CLINICAL TRIAL: NCT03849963
Title: Imaging Oxidative Metabolism and Neurotransmitter Synthesis in the Human Brain
Acronym: HP Brain
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jae Mo Park, Principal Investigator, University of Texas Southwestern Medical Center
Other Study IDs: STU-2018-0013
Record Dates: First submitted 2019-02-14; First posted 2019-02-21 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Brain Metabolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyperpolarized [13C]pyruvate: Hyperpolarized stable isotope injection ([13C]pyruvate) during magnetic resonance spectroscopic imaging

SUMMARY:
Investigators propose to develop hyperpolarized [13C]-labeled pyruvate as potential imaging probes to assess two essential in vivo processes in cerebral metabolism: oxidative metabolism and synthesis of a neurotransmitter in this observational study.

DETAILED DESCRIPTION:
Investigators will perform a pilot study to test the translational feasibility by evaluating sensitivity and repeatability of hyperpolarized [1-13C]pyruvate and [2-13C]pyruvate in healthy human subjects (n =10 each). Each subject will be imaged twice using the same hyperpolarized substrate with an interval (<45min) between the injections to evaluate repeatability. Finally, eight subjects will be imaged with both hyperpolarized [1-13C]pyruvate and [2-13C]pyruvate for comparison.

ELIGIBILITY:
Inclusion Criteria:

* 18 through 60 years of age.
* Healthy, with no neurological abnormalities.
* Ability to understand and the willingness to sign a written informed consent.
* All races and ethnicities will be included; subjects must be able to read and speak the English language.

Exclusion Criteria:

* Metallic foreign bodies on the scalp or cranium which may interfere with MRI acquisitions
* Major debilitating neurological disease including, but not limited to, stroke, CVA, dementia and tumor that would limit compliance with study requirements
* Under influence of illicit drugs which are known to alter brain physiology/metabolism including, but not limited to cocaine, lysergic acid diethylamide (LSD), and marijuana at the time of MRI/MRSI scanning.
* Under influence of antiepileptic drugs at the time of MRI/MRSI scanning.
* Any contraindication per MRI Screening Form including
* Implants contraindicated at 3T, pacemakers
* Implantable Cardioverter Defibrillator (ICD)
* Claustrophobia
* Medically unstable including
* Heart failure
* Severe left ventricular outflow tract (LVOT) obstruction
* Unstable angina
* Pregnancy
* Lactating

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of 13C ratio maps in the brain of healthy participants | Measurements made during study scan
  Product ratios (Bicarbonate/Lactate, Glutamate/Lactate) will be acquired from the hyperpolarized 13C imaging

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern - Advanced Imaging Research Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No